CLINICAL TRIAL: NCT04879888
Title: Estudio clínico Fase I de Inmunoterapia Con Vacunas sintéticas Personalizadas en Pacientes Con cáncer de Mama Triple Negativo
Brief Title: Personalized Vaccine for Cancer Immunotherapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Universidad Nacional de Colombia (Other)
Collaborators: Fundación Salud de los Andes (Other); Instituto Colombiano para el Desarrollo de la Ciencia y la Tecnología (COLCIENCIAS) (Other Government); Subred Integrada de Servicios de Salud Sur ESE - Colombia (South America) (Unknown)
Responsible Party: Principal Investigator, Carlos Alberto Parra Lopez, Full Professor, Universidad Nacional de Colombia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VP-CMTN-UN-2017
Record Dates: First submitted 2021-04-30; First posted 2021-05-10 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Breast Cancer Female
Keywords: Triple negative breast cancer; Neo-adjuvant chemotherapy; Dendritic cells; Peptide; Immunotherapy; Immune-monitoring; Personalized vaccines
MeSH Terms: conditions — Triple Negative Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vacuna (Experimental): Triple-negative breast cancer patients with specific tumor mutation, with six doses of peptide-pulsed autologous dendritic cells after surgery.
  Interventions: Biological: Peptide pulsed Dendritic cell

INTERVENTIONS:
Biological: Peptide pulsed Dendritic cell — Intradermal vaccination with peptide-pulsed autologous dendritic cells in 200 µL of patient's serum in six doses weekly after surgery.

SUMMARY:
Due to their genetic instability, breast tumors that do not express receptors for Estrogens, Progestagens or amplify the Her2 / neu oncogene [called triple-negative breast cancer (TNTC)] and other tumors such as melanoma, non-small cell lung cancer, accumulate numerous mutations that make them highly resistant to different regimens of chemo- or radiotherapy, thereby generating high morbidity and mortality. However, immunology can turn the genetic instability of tumors into the Achilles' tendon. Evidence of this has been revealed in Phase I clinical studies in patients with melanoma and lung cancer in an advanced stage of metastasis treated with Ipilimumab (anti-CTLA4) to decrease immunosuppression, in whom peptides containing mutations presented in Major Complex molecules Histocompatibility of Class I (HCM I) of the tumor itself results in their recognition as "foreign" neo-antigens leading to the efficient destruction of the tumor by anti-tumor CD8 + T lymphocytes that are amplified when they are vaccinated with these peptides.

For this reason, the identification of non-synonymous mutations of single amino acid and vaccination with 25 amino acid peptides that incorporate these mutations (synthetic vaccines) is emerging today as an alternative for immunotherapy of cancers responsible for high mortality in humans. In an approach that takes 16 weeks, today, it is possible to go from the analysis of the tumor's transcriptome (which allows identifying the universe of tumor mutations) to the patient's vaccination with a personalized vaccine that contains neo-antigens of his tumor.

TNBC is the most aggressive breast tumor, representing around 25% of breast cancers in our environment. While generally, at least 30% of women with other types of metastatic breast cancer survive 5 years after diagnosis, most patients diagnosed with metastatic CMTN die within this time. The lack of selective therapies and the poor prognosis of patients with NTMC make their therapeutic management difficult, so the implementation of new therapies for this type of tumor is the main focus of researchers who seek more effective and selective treatments to improve the life expectancy of patients without compromising their quality of life. The genetic instability and high rate of mutations of the TNBC most likely favor the generation of neo-epitopes. Still, due to the immunosuppressive environment of the tumor, it escapes the immunosurveillance of the immune system. Despite the high mortality induced by this tumor, a percentage of patients treated with neoadjuvant chemotherapy with agents such as Doxorubicin and Cyclophosphamide (AC) + Taxanes respond to this chemotherapy regimen. In particular, the anti-tumor effect of AC is attributed to two things: (i) the direct cytotoxic effect on the tumor cell, (ii) the immunostimulation of T lymphocytes promoted by Immunogenic Cell Death (ICM) selectively induced by these drugs. Therefore, in this project, we propose to carry out the first clinical study in Colombia of vaccination of patients with TNBC with synthetic peptides that contain mutations of their own tumor to evaluate the immunogenicity and safety of this type of personalized vaccine as a therapeutic alternative for this tumor. Achieving the specific objectives set out in this project would mean that we have been validated in Colombia the experimental design necessary to identify unique epitopes in tumors and demonstrate the safety and immunogenicity of these vaccines. We consider that having achieved the above; we will have taken an important step towards the implementation in our country of the use of this type of vaccine for immunotherapy not only of TNBC but of other tumors such as glioblastoma, gastric, esophagus, and pancreas, highly fatal due to its high mutation rate.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of ductal cancer who enter the primary or neoadjuvant chemotherapy regimen treated with Doxorubicin or Cyclophosphamide.
* Patients with breast cancer with the HLA-A * 02: 01 haplotype.
* Women of legal age who are not pregnant or breastfeeding (patients or controls).
* Patients who have histologically confirmed primary breast carcinoma of the ductal type.
* Karnofsky index greater than 70%
* Voluntary acceptance of informed consent.

Exclusion Criteria:

* Patients with a diagnosis of triple-negative breast cancer.
* Pregnant patients
* Patients under age or over 70 years
* Patients diagnosed with autoimmune diseases
* The patient has a Karnofsky lower than 70% or an ECOG higher than 1.
* Patients who have received some therapy as a treatment for their tumor pathology (radiotherapy, chemotherapy, immunotherapy, or gene therapy).
* Active autoimmune disease requiring treatment or a history of autoimmune disease that could be exacerbated by treatment. Patients with endocrine disease controlled by replacement therapy, including thyroid disease, adrenal disease, and vitiligo, can be included.
* Presence of a chronic or acute infection, such as HIV, viral hepatitis, or tuberculosis, before or after signing the informed consent.
* Use of immunosuppressants within 4 weeks before the trial (e.g., corticosteroids), such as azathioprine, prednisone, or cyclosporine A. The use of local steroids (topical, nasal, or inhaled) may be acceptable.
* Clinically significant cardiomyopathy, which requires treatment.
* Splenectomized patients.
* Patients who do not receive the neoadjuvant chemotherapy regimen with Doxorubicin and cyclophosphamide for three cycles or receive some other type of complementary therapy such as taxanes.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2016-12-30 (Actual); Study Completion 2017-07-30 (Actual)

PRIMARY OUTCOMES:
Number of adverse effects | From day 0 (vaccination 1) until 1 month after last vaccination
  Evaluation of number and severity of the adverse effects in the vaccinated patients

CONTACTS AND LOCATIONS:
Overall Officials: Carlos A Parra-López, MD, PhD, Principal Investigator — Full time professor
Locations (1):
- Facultad de Medicina - Universidad Nacional de Colombia, Bogota, Cundinamarca, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bernal-Estevez D, Sanchez R, Tejada RE, Parra-Lopez C. Chemotherapy and radiation therapy elicits tumor specific T cell responses in a breast cancer patient. BMC Cancer. 2016 Aug 3;16:591. doi: 10.1186/s12885-016-2625-2. PMID 27484900
- See also: Dendritic cell generation — https://symbiosisonlinepublishing.com/immunology/immunology53.php